CLINICAL TRIAL: NCT04811989
Title: Impact of Educational Interventions on Diabetic Foot Self-care: A Pragmatic Randomized Controlled Trial
Brief Title: Educational Interventions on Diabetic Foot Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Gabriela Ferreira, Principal Investigator, Master, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEICVS134/2020
Record Dates: First submitted 2021-03-14; First posted 2021-03-23 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus; Diabetic Foot
Keywords: Education; Foot care adherence; Foot health; Knowledge; Illness representations; Health literacy; Video-based intervention; Informative Leaflet
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at a ratio of 1:1 for the two conditions - Video Watching Group or Real-time Leaflet Reading Group versus Standard Care Group - into blocks of variable size, multiples of two. This randomization will be stratified according to the hospital (hospital 1 versus hospital 2) and the presence or absence of active diabetic foot ulcer.
Who Masked: Participant
Masking Description: Randomisation will be performed through an online random number generator, by a researcher external to the team of this study, to ensure the concealment of the allocation of participants by the several groups (Pandis, 2012). It will not be possible to conceal the group to which the patient was allocated to the medical and nursing team, since they have to administer the intervention or the researcher who will have to inform the respective team and administer the intervention in the Reading Group. Only the participants will be blind to the group to which they have been allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video Watching Group (Experimental): Participants will watch an instructive video on diabetic foot care and will receive face-to-face teaching on diabetic foot care.
  Interventions: Behavioral: Instructive video on diabetic foot care; Behavioral: Face-to-face teaching
- Real-time Leaflet Reading Group (Experimental): Participants will receive a leaflet with diabetic foot care information, whose reading will be guided in real-time by the Researcher, and will also receive face-to-face teaching on diabetic foot care.
  Interventions: Behavioral: Informative leaflet with real-time guided reading; Behavioral: Face-to-face teaching
- Standard Care Group (Active Comparator): Participants will receive the standard care that includes face-to-face teaching about diabetic foot care and will take a leaflet on diabetic foot care to read at home.
  Interventions: Behavioral: Informative leaflet to read at home; Behavioral: Face-to-face teaching

INTERVENTIONS:
Behavioral: Instructive video on diabetic foot care — In the video, the diabetic foot care is presented verbally and appropriately captioned, as well as exemplified by real patients and health professionals from the hospital
  Arms: Video Watching Group
Behavioral: Informative leaflet with real-time guided reading — The leaflet has information about diabetic foot care. Researcher will guide its reading with patients.
  Arms: Real-time Leaflet Reading Group
Behavioral: Informative leaflet to read at home — Patients receive a leaflet about diabetic foot care to read at home.
  Arms: Standard Care Group
Behavioral: Face-to-face teaching — Face-to-face teaching includes the teaching about diabetic foot care during the consultation by health professionals.

SUMMARY:
Diabetes mellitus currently affects 463 million people worldwide. One of the most serious complications of diabetes is the diabetic foot. Adequate foot care behaviours reduce the risk of ulcers, infections, and amputations, and improve the quality of life, in these patients.

This Pragmatic Randomized Controlled Trial aims to analyse the impact of different educational strategies - an instructive video (Video Watching Group - Experimental Group 1) compared with a leaflet on foot care with real-time guided reading (Real-Time Leaflet Reading Group - Experimental Group 2) and with standard teaching on diabetic foot care (Standard Care - Control Group) - on adherence and knowledge regarding diabetic foot care, as well as on patient's perception of their foot health. Participants will be assessed at the first consultation of the diabetic foot (T0), about two weeks after the first assessment (T1), and three months after the T0 in a follow-up assessment (T2), with T1 and T2 being performed through telephone calls, after obtaining the patients' consent.

The results of the present study will inform educational interventions regarding foot care adherence in patients with diabetic foot, in order to decrease the likelihood of developing diabetic foot ulcers and, consequently, to reduce amputation rates and the several associated costs, contributing to improving patients' quality of life.

DETAILED DESCRIPTION:
Specific Aims

1. To analyze the contribution of sociodemographic, clinical, and psychological variables to diabetic foot care adherence and knowledge, and perceived foot health, over time.
2. To analyze the differences between groups over time in diabetic foot care adherence, knowledge on foot care, and perceived foot health.
3. To examine the mediating role of representations about diabetic foot in the relationship between knowledge about foot care and adherence to diabetic foot care, over time, controlling for health literacy.
4. To examine the moderating role of foot pain, foot function, and footwear between representations about diabetic foot and adherence to diabetic foot care/ perceived foot health, over time.

Data Analysis:

Generalized Mixed Models, which allow examining changes over time including longitudinal mediation and moderation.

Sample size calculation:

Considering a dropout rate of 10%, the sample size required is 60 patients (20 per group).

Procedure:

Participants will be assessed at the first consultation of the diabetic foot (T0), about two weeks after the first assessment (T1), and three months after the T0 in a follow-up assessment (T2), with T1 and T2 being performed through telephone calls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Diabetes mellitus;
* Diagnosis of Diabetic Foot;
* To benefit from the first assessment and follow-up at the Multidisciplinary Diabetic Foot Consultation of the hospitals where data collection will take place.

Exclusion Criteria:

* Presence of clinical dementia described in the patient's clinical record;
* Cognitive disability to answer the questionnaires;
* Severe visual and/or hearing impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Adherence to the diabetic foot care behaviours | Changes from baseline to two weeks post-test and after a three month follow-up
  Adherence to foot care behaviors will be assessed through the Nottingham Assessment of Functional Foot Care (Lincoln, Jeffcoate, Ince, Smith, & Radford, 2007). Composed of 29 items whose answers are given on a Likert scale ranging from 0 to 3. Higher scores correspond to a higher frequency of foot care behaviors.
Adherence to the diabetic foot care behaviours | Changes from baseline to two weeks post-test and after a three month follow-up
  The level of foot self-care (indirect measure of adherence) will be assessed through the subscale of Foot Care of the Summary Diabetes Self-Care Activities Questionnaire (Original Version by Toobert, Hampson, & Glasgow, 2000; Portuguese Version by Bastos, Severo, & Lopes, 2007). Composed of 3 items in which patients are asked how many of the last seven days did they perform the respective foot care behaviour. Therefore, answers are given on a scale between 0 and 7, and its score is calculated through the mean number of days. Higher scores indicate higher levels of foot self-care.
Knowledge on foot care | Changes from baseline to two weeks post-test and after a three month follow-up
  Knowledge on foot care will be assessed through the Questionnaire on Knowledge of Foot Care (Hasnain & Sheikh, 2009). Each correct answer is scored with 1 point and higher scores indicate better knowledge about foot care.
General foot health | Changes from baseline to two weeks post-test and after a three month follow-up
  General foot health will be assessed through the respective subscale of the Foot Health Status Questionnaire (FHSQ; Bennett, Patterson, Wearing, & Baglioni, 1998). Scores are transformed into a scale of 0 to 100, where 0 corresponds to the perception of poor foot health state/condition and 100 to the perception of excellent foot health.

SECONDARY OUTCOMES:
Representations about diabetic foot | Changes from baseline to two weeks post-test and after a three month follow-up
  Representations about diabetic foot will be assessed through the Illness Perception Questionnaire - Brief (IPQ-B; Figueiras et al., 2010). The response scale ranges from 0 to 10. Higher scores indicate more threatening representations regarding diabetic foot.

OTHER OUTCOMES:
Foot pain | Baseline (T0), two weeks post-test (T1), three months follow-up (T2)
  Foot pain will be assessed through the respective subscale of the Foot Health Status Questionnaire (Bennett, Patterson, Wearing, & Baglioni, 1998). Scores are transformed into a scale of 0 to 100, where 0 corresponds to significant or extreme foot pain and 100 to no foot pain or discomfort.
Foot function | Baseline (T0), two weeks post-test (T1), three months follow-up (T2)
  Foot function will be assessed through the respective subscale of the Foot Health Status Questionnaire (FHSQ; Bennett, Patterson, Wearing, & Baglioni, 1998). Scores are transformed into a scale of 0 to 100, where 0 corresponds to severe limitation in the performance of physical activities because of the feet and 100 to no limitation.
Footwear | Baseline (T0), two weeks post-test (T1), three months follow-up (T2)
  Footwear will be assessed through the respective subscale of the Foot Health Status Questionnaire (FHSQ; Bennett, Patterson, Wearing, & Baglioni, 1998). Scores are transformed into a scale of 0 to 100, where 0 corresponds to severe problems obtaining appropriate footwear and 100 to no problems.
Clinical Data | Baseline (T0)
  Clinical variables (e.g., HbA1c levels, presence/absence of active ulcer and duration of diabetic foot ulcer, recommendation to use therapeutic footwear) will be assessed through a Clinical Questionnaire developed for this study
Health literacy | Baseline (T0)
  Health literacy will be assessed through the Medical Term Recognition Test (METER; Paiva et al., 2014).
Sociodemographic data | Baseline (T0)
  The sample will be characterized using a Sociodemographic Questionnaire developed for this study (e.g. age, marital status, gender, socio-economic level).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Ferreira, Master, Principal Investigator — School of Psychology, University of Minho
Locations (2):
- Portugal (2):
  - Clínica do Pé Diabético, Centro Hospitalar do Tâmega e Sousa, Penafiel, Porto District
  - Centro Hospitalar Universitário do Porto, Porto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bastos F, Severo M, Lopes C. [Psychometric analysis of diabetes self-care scale (translated and adapted to Portuguese)]. Acta Med Port. 2007 Jan-Feb;20(1):11-20. Epub 2007 May 23. Portuguese. PMID 17624279
- [Background] Bennett PJ, Patterson C, Wearing S, Baglioni T. Development and validation of a questionnaire designed to measure foot-health status. J Am Podiatr Med Assoc. 1998 Sep;88(9):419-28. doi: 10.7547/87507315-88-9-419. PMID 9770933
- [Background] Figueiras M, Marcelino DS, Claudino A, Cortes MA, Maroco J, Weinman J. Patients' illness schemata of hypertension: the role of beliefs for the choice of treatment. Psychol Health. 2010 Apr;25(4):507-17. doi: 10.1080/08870440802578961. PMID 20204931
- [Background] Hasnain S, Sheikh NH. Knowledge and practices regarding foot care in diabetic patients visiting diabetic clinic in Jinnah Hospital, Lahore. J Pak Med Assoc. 2009 Oct;59(10):687-90. PMID 19813683
- [Background] Lincoln, N. B., Jeffcoate, W. J., Ince, P., Smith, M., & Radford, K. A. (2007). Validation of a new measure of protective footcare behaviour: the Nottingham Assessment of Functional Footcare (NAFF). Practical Diabetes International, 24, 207-211. doi:10.1002/pdi.1099
- [Background] Paiva D, Silva S, Severo M, Ferreira P, Santos O, Lunet N, Azevedo A. Cross-cultural adaptation and validation of the health literacy assessment tool METER in the Portuguese adult population. Patient Educ Couns. 2014 Nov;97(2):269-75. doi: 10.1016/j.pec.2014.07.024. Epub 2014 Jul 22. PMID 25107513
- [Background] Pandis N. Randomization. Part 3: allocation concealment and randomization implementation. Am J Orthod Dentofacial Orthop. 2012 Jan;141(1):126-8. doi: 10.1016/j.ajodo.2011.09.003. No abstract available. PMID 22196195
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844